CLINICAL TRIAL: NCT03078062
Title: Impact of Intravenous Dexamethasone on the Duration of Sensory and Motor Block Following a Bupivacaine-based Spinal Anesthesia
Brief Title: Impact of Dexamethasone on the Duration of Sensory and Motor Block Following Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16.374
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Spinal Anesthesia; Prolonged Sensory Block; Prolonged Motor Block
Keywords: Spinal anesthesia; Motor block; Sensory block; Dexamethasone
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients in both groups will receive the study drug (dexamethasone or placebo) in the same volume of normal saline. The study drug will be prepared by an independent assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): During the performance of spinal anesthesia using isobaric 0.5% bupivacaine 12 mg, an intravenous infusion of dexamethasone 8 mg (2 ml) will be initiated. The study drug will be administered over 5 -10 minutes diluted in a 500 ml bag of Normal Saline for a total volume of 502 ml. The study drug will be prepared by an independent assistant.
  Interventions: Drug: Dexamethasone
- Normal Saline (Placebo Comparator): During the performance of spinal anesthesia using isobaric 0.5% bupivacaine 12 mg, an intravenous infusion of 502 ml of Normal Saline will be initiated. The infusion will be administered over 5 -10 minutes. The study drug will be prepared by an independent assistant.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Administration of a single-dose of intravenous dexamethasone 8 mg during spinal anesthesia
  Other Names: Decadron
  Arms: Dexamethasone
Drug: Normal saline — Administration of a single-dose of Normal saline during spinal anesthesia
  Other Names: Placebo
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to assess the effect of a single-dose of intravenous dexamethasone 8 mg on the duration of sensory and motor blockade following spinal anesthesia with isobaric bupivacaine.

The hypothesis of the study is that intravenous dexamethasone will significantly prolong (by more than 20 minutes) the duration of spinal anesthesia.

DETAILED DESCRIPTION:
Spinal anesthesia is commonly used for lower body surgery. The injection of local anesthetics in the lumbar intrathecal space allows the desensitization of the lower body by blocking sensory and motor nerve roots. In return, spinal anesthesia causes a sympathetic block which is associated with deleterious hemodynamic effects such as hypotension.

Using intravenous or intrathecal adjuvants to local anesthetics may prolong the duration of sensory and motor blockade following spinal anesthesia. Various intrathecal additives have been studied such as opioids, adrenalin, clonidine, dexmedetomidine, midazolam, ketamine, magnesium, ketorolac and neostigmine. Most of them failed to prolong the duration of spinal anesthesia and side-effects have restricted their use.

Dexamethasone is a potent corticosteroid with a half-life of 36 to 72 hours and an onset of action of 1 to 2 hours. The safety of single doses of intravenous dexamethasone is well documented. Dexamethasone is widely used in anesthesia to prevent nausea and vomiting and treat post-extubation sore throat and postoperative shivering. It is also increasingly used in orthopaedic surgery to reduce opioid needs without increasing the risks of infection, wound dehiscence and osteonecrosis. The use of dexamethasone in the perioperative period reduces postoperative edema allowing early mobilization and improved functional recovery.

Recent studies have demonstrated that both perineural and intrathecal administration of dexamethasone can prolong the duration of peripheral and spinal anesthesia. However, dexamethasone has not been approved by health authorities for these indications and thus, the safety of this practice remains controversial. A recent study has compared peripheral to intravenous administration of dexamethasone for interscalene blocks. This study demonstrated the equivalency of these regimens in increasing the analgesic duration of a single-shot interscalene block.

The impact of intravenous dexamethasone on the duration of spinal anesthesia remains unknown. This study will investigate the effect of a single-dose of dexamethasone 8 mg on the duration of the sensory and motor block following spinal anesthesia.

Sixty patients scheduled for lower body surgery under spinal anesthesia will be considered for this study.

After placement of standard non-invasive monitoring, spinal anesthesia will be performed in the sitting position using a 25 gauge (GA) pencil point needle (Whitacre, Pencan). After aspiration of cerebrospinal fluid (CSF), a dose of isobaric 0.5% bupivacaine 12 mg will be injected. The aspiration of CSF will be repeated at the end of the injection. While performing spinal anesthesia, an intravenous infusion of dexamethasone 8 mg or placebo will be initiated according to randomization.

Subsequently, the patient will be placed in supine position. Sensory block will be measured by loss of sensation to pinprick at 5, 10, 20 and 30 minutes following spinal anesthesia and then every 15 minutes until confirmation of regression by two dermatomes. Loss of sensation will be assessed every 30 minutes thereafter. Motor block will be assessed using the Bromage scale at the same frequency until full recovery.

Sedation will be allowed during the performance of the spinal anesthesia technique and surgery. In case of unsatisfactory quality of spinal anesthesia, general anesthesia will be performed.

At the end of surgery, patients will be transferred to the recovery room. Multimodal analgesia including celecoxib and acetaminophen will be administered. Pain will be assessed using a verbal numeric pain scale (VNPS) of 0 to 10, where 0 means "No pain" and 10 means "Worst pain imaginable". Intravenous hydromorphone will be administered when VNPS is superior to 3. Postoperative nausea and vomiting will be managed with intravenous ondansetron, dimenhydrinate and haloperidol.

Opioid intake, presence of side-effects and quality of sleep will be assessed during the first 24 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lower body surgery under spinal anesthesia
* American Society of Anesthesiologists' physical status of 1 to 3

Exclusion Criteria:

* Contraindication to spinal anesthesia (coagulopathy, local infection at the site of injection)
* Pre-existing neuropathy or nerve block that could compromise study assessments
* Preoperative use of systemic corticosteroids
* Allergy or hypersensitivity to local anesthetics, dexamethasone or other drugs used in this study
* Patient refusal or inability to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Regression of sensory block by 2 dermatomes | At regression of spinal anesthesia by 2 dermatomes, approximately 2 hours after surgery
  Loss of pinprick sensation by Von Frey filaments from the injection of bupivacaine for spinal anesthesia until regression of the sensory block by two dermatomes from the peak sensory level

SECONDARY OUTCOMES:
Duration of motor block | At 5,10, 20 and 30 minutes following spinal anesthesia, then every 15 minutes until regression of 2 dermatomes and every 30 minutes thereafter until complete recovery, approximately 4 hours after surgery
  Using the Bromage scale from the time of injection of bupivacaine for spinal anesthesia until complete recovery of motor block
Onset of sensory block | Up to 30 minutes following spinal anesthesia
  Time from injection of bupivacaine for spinal anesthesia to reduction of sensitivity using loss of pinprick sensation
Onset of motor block | Up to 30 minutes following spinal anesthesia
  Time from injection of bupivacaine for spinal anesthesia to reduction of lower limbs movement using the Bromage scale
Quality of motor block | Up to 30 minutes following spinal anesthesia
  Maximal Bromage score
Surgeon's satisfaction towards spinal anesthesia | At the end of surgery, on the day of randomization
  Unsatisfied or satisfied
Time to first analgesic request | From the end of surgery up to approximately six hours after surgery, on the day of randomization
  First request by the patient for an analgesic or pain superior to 3 on a scale from 0 to 10; where 0 means "no pain at all" and 10 means "worst pain imaginable"
Opioid consumption | At recovery room discharge, approximately one hour after the end of surgery on the day of randomization and 24 hours following surgery
  Total dose of opioids
Incidence of hypotension | From injection of bupivacaine for spinal anesthesia to 24 hours after surgery
  Systolic blood pressure lower than 90 mm Hg
Incidence of bradycardia | From injection of bupivacaine for spinal anesthesia to 24 hours after surgery
  Heart rate slower than 50 beats per minute
Incidence of nausea | From injection of bupivacaine for spinal anesthesia to 24 hours after surgery
  Any episode of nausea reported by the patient or nursing team
Incidence of vomiting | From injection of bupivacaine for spinal anesthesia to 24 hours after surgery
  Any episode of retching or vomiting reported by the patient or nursing team
Incidence of urinary retention | From injection of bupivacaine for spinal anesthesia to 24 hours after surgery
  Any episode of urinary retention reported by the patient or nursing team
Incidence of shivering | From injection of bupivacaine for spinal anesthesia to 24 hours after surgery
  Any episode of shivering reported by the patient or nursing team
Incidence of headache | From injection of bupivacaine for spinal anesthesia to 24 hours after surgery
  Any episode of headache reported by the patient or nursing team
Quality of sleep | At 24 hours after surgery
  Described by the patient as good or bad
Duration of sensory block | At 5,10, 20 and 30 minutes following spinal anesthesia, then every 15 minutes until regression by 2 dermatomes and every 30 minutes thereafter until complete recovery, approximately 4 hours after surgery
  Loss of pinprick sensation by Von Frey filaments from the injection of bupivacaine for spinal anesthesia until complete recovery

CONTACTS AND LOCATIONS:
Overall Officials: Stephan R Williams, Md, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No